CLINICAL TRIAL: NCT03123965
Title: Expanded Access to Glecaprevir/ Pibrentasvir
Status: Approved for marketing | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C16-563
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis C Virus Infection
Keywords: Special Access Scheme; Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir; pibrentasvir

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: glecaprevir — Glecaprevir will be administered orally.
  Other Names: ABT-493
Drug: pibrentasvir — Pibrentasvir will be administered orally.
  Other Names: ABT-530

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to glecaprevir/ pibrentasvir prior to approval by the local regulatory agency. Availability will depend on territory eligibility. Participating sites will be added as they apply for and are approved for the EAP. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (1):
- Univ Medical Ctr Ljubljana /ID# 161419, Ljubljana, Slovenia